CLINICAL TRIAL: NCT06763978
Title: Comparative Analysis of Isolated Venous, Isolated Arterial, and Standard Access for Transcatheter Closure of Patent Ductus Arteriosus (PDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Nouran Mostafa Mansour, DR., Egyptian Biomedical Research Network
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 36264PR897/10/24
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Hemodynamically Significant PDA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 152 patients who underwent ordinary transcatheter closure technique using both arterial and venous a (Active Comparator)
  Interventions: Device: Transcatheter PDA closure
- 113 patients who underwent transcatheter closure using exclusive venous access only. (Active Comparator)
  Interventions: Device: Transcatheter PDA closure
- included 92 patients who underwent transcatheter closure using exclusive arterial access only. (Active Comparator)
  Interventions: Device: Transcatheter PDA closure

INTERVENTIONS:
Device: Transcatheter PDA closure — Transcatheter PDA closure

SUMMARY:
We enrolled all patients with a hemodynamically significant PDA demonstrated by patient clinical condition, and by PDA size & left chamber dilatation on echocardiography attending at Cardiology Department to we compare the use of a single venous access and a single arterial access with the standard approach requiring both venous and arterial access for transcatheter PDA closure regarding the outcome & complications.

ELIGIBILITY:
Inclusion Criteria:

* any patient with hemodynamically significant PDA

Exclusion Criteria:

* patient with pulmonary hypertension and Eisenmenger syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
procedural and fluoroscopy time | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No